CLINICAL TRIAL: NCT00665626
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Dose Study of R935788 in Patients With Rheumatoid Arthritis Who Have Failed at Least One Biologic
Brief Title: Efficacy and Safety Study of R935788 Tablets to Treat Rheumatoid Arthritis (Taski-3)
Acronym: Taski-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-935788-011
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Results first posted 2016-07-15 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Fostamatinib disodium (R935788) 100 mg tablet, orally, twice-a-day
  Interventions: Drug: Fostamatinib disodium (R935788)
- Arm 2 (Placebo Comparator): Placebo, orally, twice-a-day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fostamatinib disodium (R935788) — R935788 100 mg tablet, orally, twice-a-day
  Arms: Arm 1
Drug: Placebo — Placebo, orally, twice-a-day
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine whether the Spleen Tyrosine Kinase (Syk) Inhibitor, R935788 (R788) at a dose of 100 mg, tablet, orally, twice-a-day is effective in the treatment of Rheumatoid Arthritis in patients who have 'failed' a biologic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent by signing an IRB/EC-approved Informed Consent Form (ICF) prior to admission to this study.
* Males and females, 18 years of age or older, with active RA for at least 12 months prior to Day 1 dosing
* Are currently receiving or previously had received a biologic therapy with an inhibitor of TNF, rituximab, abatacept, or anakinra at an approved labeled dose for ≥3 months prior to Day 1 dosing and are designated as biologic therapy failures for lack of efficacy, safety, or tolerability.
* Patients may receive stable doses of methotrexate (MTX), azathioprine (not in combination with MTX), leflunomide (not in combination with MTX), sulfasalazine, chloroquine, hydroxychloroquine, gold, NSAIDs (including COX2 inhibitors), minocycline, or doxycycline. The dose must have been stable for at least 30 days prior to Day 1 dosing and must not be changed during the washout, screening and treatment periods, unless dictated by tolerability requirements. Patients who are taking MTX must have been receiving weekly MTX doses (7.5-25 mg/week) for a minimum of 3 months prior to Day 1 dosing and must be receiving a stable MTX dose, with no change in route, for the previous 6 weeks prior to Day 1 dosing. Patients who are receiving MTX must also be receiving folic or folinic acid supplementation at a stable dose for at least 6 weeks prior to Day 1 dosing.
* Females of childbearing potential must be fully informed of the potential for R788 to adversely affect the fetus and, if sexually active, must agree to use a well established method of birth control during the study (oral contraceptive, mechanical barrier, long acting hormonal agent). These patients must not be lactating and must have a negative urine pregnancy test at the time of randomization and at each laboratory determination.
* The patient must otherwise be in good health as determined by the Investigator on the basis of medical history, physical examination, and laboratory screening tests during the screening period. See exclusion criteria for specific exclusions.
* In the Investigator's opinion, the patient has the ability to understand the nature of the study and any hazards of participation, and to communicate satisfactorily with the Investigator and to participate in, and to comply with, the requirements of the entire protocol.

Exclusion Criteria:

* The patient has a history of, or a concurrent, clinically significant illness, medical condition (other than arthritis) or laboratory abnormality that, in the Investigator's opinion, could affect the conduct of the study. Specifically, excluded are patients with the following:

  1. uncontrolled or poorly controlled hypertension;
  2. other autoimmune disease (psoriatic arthritis, lupus, mixed connective disorder) or arthritis syndromes (gout, Lyme disease, Reiter's syndrome);
  3. recent serious surgery or infectious disease;
  4. recent history ( of, or treatment for, a malignancy other than nonmelanomatous skin cancer, or any history of lymphoma;
  5. Hepatitis B;
  6. Hepatitis C;
  7. interstitial pneumonitis or active pulmonary infection on chest x-ray
  8. Tuberculosis (TB)
  9. known laboratory abnormalities
* The patient has a history of substance abuse, drug addiction or alcoholism. Patients may consume up to 4 units of alcohol per week; however, alcohol should be avoided in the 72 hours prior to lab assessments. Patients who cannot reliably comply with this should be excluded. A unit of alcohol is defined as the following: Beer=12 oz or 355 mL; wine = 5 oz or 148 mL; sweet dessert wine=3 oz or 89 mL; 80 proof distilled spirits= 1.5 oz or 44 mL.
* The patient has been treated previously treated with R788 under a different protocol.
* The patient has a pacemaker, aneurysm clip or other contraindication to MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Magilavy, MD, Study Director — Rigel Pharmaceuticals
Locations (44):
- United States (27):
  - Arthritis & Rheumatic Disease Specialties, Aventura, California
  - Desert Medical Advances, Palm Desert, California
  - San Diego Arthritis & Medical Clinic, San Diego, California
  - Department of Rheumatology, Washington D.C., District of Columbia
  - RASF-Clinical Research Center, Boca Raton, Florida
  - Florida Medical Research Institute, Gainsville, Florida
  - Paddock Park Clinical Research, Ocala, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - Intermountain Orthopedics, Boise, Idaho
  - Rheumatology Associates, SC, Chicago, Illinois
  - Memorial Medical Group Clinical Research Inst, South Bend, Indiana
  - Center for Arthritis & Osteoperosis, Elizabethtown, Kentucky
  - The Osteoporosis & Clinical Trials Center, Cumberland, Maryland
  - The Osteoporosis & Clinical Trials Center, Hagerstown, Maryland
  - Fiechtner Research, Inc., Lansing, Michigan
  - Westroads Medical Group, Omaha, Nebraska
  - North Shore Long Island Jewich Health System, Lake Success, New York
  - Andrew Porges, MD PC, Roslyn, New York
  - Rheumatology Associates of Long Island, Smithtown, New York
  - Clinical Research Division, Mayfield Village, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Rheumatology Associates, Erie, Pennsylvania
  - Clinical Research Center of Reading, LLP, West Reading, Pennsylvania
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - Austin Rheumatology & Research, Austin, Texas
  - Houston Institute for Clinical Research, Houston, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
- Belgium (3):
  - ZNA Middelheim, Antwepen
  - UZ Gent, Ghent
  - CHU Liege, Liège
- Colombia (5):
  - Reumalab S.A., Medellín, Antioquia
  - Reumatologos del Caribe, Barranquilla, Atlántico
  - CIREEM, Bogota, Cundinamarca
  - Dr. Renato Guzman, Bogota, Cundinamarca
  - Riesgo de Fractura S.A., Bogota, Cundinamarca
- Hopital Pellegrin, Bordeaux, France
- Germany (5):
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Klinikum Eilbek, Hamburg
  - ClinPharm International GmbH Leipzig, Leipzig
  - Rheumazentrum am Universitatsklinikum Leipzig, Leipzig
  - Universitatsklinikum Wurzburg, Würzburg
- Italy (2):
  - Reumatologia Azienda Ospedaliera Universitaria, Siena
  - Azienda Ospedaliera Santa Maria della Miseri, Udine
- Instituto de Ginecologia y Reproduccion, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant received the first dose of study drug on 28 May 2008; the last participant completed the study on 09 June 2009. Participants were recruited from centers in the United States, Europe and Latin America.
Pre-assignment Details: Male/female participants who had active rheumatoid arthritis (RA) for a minimum of 12 months and who had failed prior biologic therapy were randomly assigned to receive R788 100 mg twice daily or placebo. It was planned to randomize approximately 195 participants.
Groups:
- Placebo: Placebo to R788, oral tablets, twice daily, double-blind
- R788 100 mg Bid: R788 100 mg, oral tablets, twice daily, double-blind
Period: Overall Study
Arm/Group | Placebo | R788 100 mg Bid
Started | 73 (Participants randomized) | 146 (Participants randomized)
Completed | 63 (Participants completed the study) | 124 (Participants completed the study)
Not Completed | 10 | 22
Not completed — Lack of Efficacy | 8 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Adverse Event | 1 | 9
Not completed — Due to exclusion criteria | 0 | 1
Not completed — Did not fulfil inclusion criteria | 0 | 1
Not completed — Unably to comply with dosing regimen | 0 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | R788 100 mg Bid | Total
Number analyzed (Participants) | 73 | 146 | 219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (12.29) | 56.0 (11.45) | 56.0 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 117 | 176
  Male | 14 | 29 | 43

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20 (ACR20) Response at 3 Months
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, Health Assessment Questionnaire-Disability Index (HAQ-DI); and CRP or ESR, after 3 months
Time Frame: 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Groups:
- Arm 1 - Placebo: Placebo to R788, oral tablets, twice daily, double-blind
- Arm 2 - R788 100 mg Bid: R788 100 mg, oral tablets, twice daily, double-blind
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 27 | 56

2. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 3 Months
Description: The number of participants with greater than or equal to 50% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and CRP or ESR, whichever was elevated at baseline, after 3 months
Time Frame: 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 9 | 32

3. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 3 Months
Description: The number of participants with greater than or equal to 70% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and CRP or ESR, whichever was elevated at baseline, after 3 months
Time Frame: 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 4 | 13

4. Secondary Outcome: American College of Rheumatology Index of Improvement (ACRn) at 3 Months
Description: The index of improvement in RA, where 0 indicates no improvement and 100 indicates a 100% improvement across all signs and symptoms of RA after 3 months of treatment
Time Frame: 3 months
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 63 | 124
Score | 19.85 (25.604) | 25.95 (28.624)

5. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <2.6 at 3 Months
Description: Number of participants with DAS28-CRP (measuring RA symptoms including: tender joint count, swollen joint count, patient's assessment of disease activity, and CRP in patients with high CRP at baseline), of less than 2.6. The DAS runs from 0 to 10 - higher scores indicate worse symptoms. A score of less than 2.6 indicates remission of RA symptoms
Time Frame: 3 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 41 | 88
Participants | 1 | 11

6. Secondary Outcome: Disease Activity Score-C-Reactive Protein (DAS28-CRP) <3.2 at 3 Months
Description: Number of participants with DAS28-CRP (measuring RA symptoms including: tender joint count, swollen joint count, patient's assessment of disease activity, and CRP in patients with high CRP at baseline), of less than 3.2. The DAS runs from 0 to 10 - higher scores indicate worse symptoms. A score of less than 3.2 indicates low disease activity.
Time Frame: 3 months
Population: Intent-to-Treat Population with CRP as Primary Phase Reactant
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 41 | 88
Participants | 4 | 21

7. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <2.6 at 3 Months
Description: Number of participants with DAS28-ESR (measuring RA symptoms including: tender joint count, swollen joint count, patient's assessment of disease activity, and ESR in patients with high ESR at baseline), of less than 2.6. The DAS runs from 0 to 10 - higher scores indicate worse symptoms. A score of less than 2.6 indicates remission of RA symptoms
Time Frame: 3 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 21 | 36
Participants | 5 | 4

8. Secondary Outcome: Disease Activity Score-Erythrocyte Sedimentation Rate (DAS28-ESR) <3.2 at 3 Months
Description: Number of participants with DAS28-ESR (measuring RA symptoms including: tender joint count, swollen joint count, patient's assessment of disease activity, and ESR in patients with high ESR at baseline), of less than 3.2. The DAS runs from 0 to 10 - higher scores indicate worse symptoms. A score of less than 3.2 indicates low disease activity.
Time Frame: 3 months
Population: Intent-to-Treat Population with ESR as Primary Phase Reactant
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 21 | 36
Participants | 7 | 6

9. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at Week 1
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and CRP or ESR, whichever was elevated at baseline, after 1 week.
Time Frame: 1 week
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 12 | 41

10. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at Week 2
Description: The number of participants with greater than or equal to 20% improvement in tender and swollen joint counts, AND in any 3 of the following: physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, HAQ-DI; and CRP or ESR, whichever was elevated at baseline, after 2 weeks
Time Frame: 2 weeks
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 14 | 44

11. Secondary Outcome: Rheumatoid Arthritis Magnetic Resonance Imaging Scoring (RAMRIS) Erosion Score at 3 Months
Description: Change from baseline in RAMRIS erosion score (a measure of bone erosion in the hands and wrists), calculated as the score at 3 months minus the score at baseline. The erosion score runs from 0 to 250 with lower values indicating a better clinical condition. A negative change indicates an improvement in symptoms.
Time Frame: Baseline to 3 months
Population: Intent-to-treat population with available data and received study drug. The discrepancy in the lower number of subjects than those in the ITT population is because 43 subjects either never had a complete set of MRIs (pre and post-study) or had uninterpretable results.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 60 | 115
Score | 0.94 (1.740) | 0.78 (2.174)

12. Secondary Outcome: Rheumatoid Arthritis Magnetic Resonance Imaging Scoring (RAMRIS) Osteitis Score at 3 Months
Description: Change from baseline in RAMRIS osteitis score (a measure of bone inflammation in the hands and wrists), calculated as the score at 3 months minus the score at baseline. The osteitis score runs from 0 to 75 with lower values indicating a better clinical condition. A negative change indicates an improvement in symptoms.
Time Frame: Baseline to 3 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 60 | 115
Score | 1.17 (4.848) | -0.19 (5.340)

13. Secondary Outcome: Rheumatoid Arthritis Magnetic Resonance Imaging Scoring (RAMRIS) Synovitis Score at 3 Months
Description: Change from baseline in RAMRIS synovitis score (a measure of inflammation in the joints of the hands and wrists), calculated as the score at 3 months minus the score at baseline. The synovitis score runs from 0 to 24 with lower values indicating a better clinical condition. A negative change indicates an improvement in symptoms.
Time Frame: Baseline to 3 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 60 | 115
Score | 0.35 (1.791) | -0.52 (2.499)

14. Secondary Outcome: Alanine Aminotransferase (ALT) >1.5x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 1.5 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 8 | 14

15. Secondary Outcome: Alanine Aminotransferase (ALT) >1.5-2x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 1.5 to 2 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 7 | 7

16. Secondary Outcome: Alanine Aminotransferase (ALT) >2-3x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 2 to 3 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 1 | 1

17. Secondary Outcome: Alanine Aminotransferase (ALT) >3x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 3 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 0 | 6

18. Secondary Outcome: Alanine Aminotransferase (ALT) >3-5x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 3 to 5 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 0 | 1

19. Secondary Outcome: Alanine Aminotransferase (ALT) >5-10x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 5 to 10 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 0 | 1

20. Secondary Outcome: Alanine Aminotransferase (ALT) >10x Upper Limit of Normal (ULN)
Description: The number of participants with ALT (a test of liver function) values greater than 10 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 0 | 4

21. Secondary Outcome: Aspartate Aminotransferase (AST) >1.5x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 1.5 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 4 | 11

22. Secondary Outcome: Aspartate Aminotransferase (AST) >1.5-2x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 1.5 to 2 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 3 | 4

23. Secondary Outcome: Aspartate Aminotransferase (AST) >2-3x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 2 to 3 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 0 | 2

24. Secondary Outcome: Aspartate Aminotransferase (AST) >3x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 3 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 1 | 5

25. Secondary Outcome: Aspartate Aminotransferase (AST) >3-5x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 3 to 5 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 1 | 1

26. Secondary Outcome: Aspartate Aminotransferase (AST) >5-10x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 5 to 10 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 0 | 3

27. Secondary Outcome: Aspartate Aminotransferase (AST) >10x Upper Limit of Normal (ULN)
Description: The number of participants with AST (a test of liver function) values greater than 10 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 0 | 1

28. Secondary Outcome: Alkaline Phosphatase >1.5x Upper Limit of Normal (ULN) and >1.5x Baseline
Description: The number of participants with alkaline phosphatase (a test of liver function) values greater than 1.5 times the ULN and greater than 1.5 times baseline
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 0 | 2

29. Secondary Outcome: Bilirubin >1.5x Upper Limit of Normal (ULN)
Description: The number of participants with bilirubin (a test of liver function) values greater than 1.5 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 0 | 3

30. Secondary Outcome: Bilirubin >2x Upper Limit of Normal (ULN)
Description: The number of participants with bilirubin (a test of liver function) values greater than 2 times the ULN
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 0 | 1

31. Secondary Outcome: Absolute Neutrophil Count (ANC) <1500/mm3
Description: The number of participants with ANC values less than 1500/mm3
Time Frame: Any time between baseline and 3 months
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - R788 100 mg Bid
Number analyzed (Participants) | 73 | 146
Participants | 0 | 9

ADVERSE EVENTS:
Arm/Group | Placebo | R788 100 mg Bid
Serious Adverse Events (participants affected / at risk) | 1/73 | 13/146
Other Adverse Events (participants affected / at risk) | 20/73 | 74/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | R788 100 mg Bid (N=146)
Coronary Artery Stenosis (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | R788 100 mg Bid (N=146)
Neutropenia (Blood and lymphatic system disorders) | 0 | 8
Diarrhoea (Gastrointestinal disorders) | 5 | 17
Nausea (Gastrointestinal disorders) | 2 | 13
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 9
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 12
Transaminases Increased (Investigations) | 0 | 8
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 | 1
Headache (Nervous system disorders) | 2 | 14
Hypertension (Vascular disorders) | 3 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less